CLINICAL TRIAL: NCT00755560
Title: Treatment of Asymptomatic Toxocariasis With Albendazole in Children. A Prospective, Randomized, Placebo-controlled Clinical Trial
Brief Title: Treatment of Asymptomatic Toxocariasis With Albendazole in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hospital de Niños R. Gutierrez de Buenos Aires (Other)
Responsible Party: Principal Investigator, Dr Jaime Altcheh, Service Head, Parasitology and Chagas Service, Hospital de Niños R. Gutierrez de Buenos Aires
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TOXOCARA-ALBENDAZOLE
Record Dates: First submitted 2008-09-17; First posted 2008-09-19 (Estimated); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Toxocariasis
Keywords: Toxocara; Pediatrics; Albendazole; eosinophilia; parasitology; pediatric clinical pharmacology
MeSH Terms: conditions — Toxocariasis; Eosinophilia | interventions — Albendazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Albendazole (Active Comparator): Albendazole 10 - 15 mg/kg/day BID for 15 days
  Interventions: Drug: Albendazole
- Placebo (Placebo Comparator): Placebo BID for 15 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Albendazole — Albendazole 10 - 15 mg/kg/day BID for 15 days
  Arms: Albendazole
Drug: Placebo — Placebo BID for 15 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate effectiveness of albendazole in the treatment of the asymptomatic infection with the parasite Toxocara in children. Treatment response is defined as a reduction in the number of eosinophils in blood. The study drug will be compared to placebo and randomly assigned in a double blind manner. Follow up will be prospective. 50 children (25 per group) will be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric ambulatory patients with asymptomatic toxocariasis
* Children 2 - 15 years old
* Absolute eosinophil count > 1100 / mm3
* Normal ophthalmoscopy

Exclusion Criteria:

* Treatment with a benzimidazole in the previous year
* Infection by other nematodes (Ascaris lumbricoides, strongyloides stercoralis, uncinarias, Trichuris trichuria)
* Symptomatic patients (prolonged fever, acute pneumonitis, hepatomegaly, splenomegaly, ocular compromise due to toxocara)
* Concomitant diseases
* Immunocompromised patients
* Altered liver or kidney function
* Pregnancy

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2008-09; Primary Completion 2015-07 (Actual); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Mean absolute reduction in eosinophil count from baseline | 12 months after treatment

SECONDARY OUTCOMES:
Reduction in eosinophil count in more than 60% from baseline | 1 year
Incidence of adverse drug events | 3, 6, 9 and 12 months after treatment
Mean absolute reduction in eosinophil count | 3, 6, 9 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Altcheh, MD, Study Chair — Parasitology Division, Children's Hospital "R Gutierrez" of Buenos Aires; Hector Freilij, MD, Principal Investigator — Parasitology Division, Children's Hospital "R Gutierrez" of Buenos Aires
Locations (1):
- Parasitology Division, Children's Hospital "R Gutierrez" of Buenos Aires, Buenos Aires, Argentina

IPD SHARING:
Plan to Share IPD: Undecided